CLINICAL TRIAL: NCT00367367
Title: Endometrial Hysteroscopy and Curettage Prior to Embryo Transfer
Brief Title: Endometrial Curettage Before Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3280105; Ministry of Heath:920050038; Genetics committee: 2005-061
Record Dates: First submitted 2006-08-20; First posted 2006-08-22 (Estimated); Last update posted 2006-08-22 (Estimated); Status verified 2006-08

CONDITIONS: Infertility
Keywords: embryo transfer; hysteroscopy; curettage; iv-vitro fertilization; molecular markers; endometrial receptivity; endometrial dating
MeSH Terms: conditions — Infertility | interventions — Hysteroscopy; Curettage

INTERVENTIONS:
Procedure: Hysteroscopy and Curettage

SUMMARY:
Studies have shown that endometrial sampling in the month prior to embryo transfer may increase pregnancy rates. We wish to test this hypothesis by performing a hysteroscopy and curettage in the month proceeding embryo transfer during IVF, IVF/ICSI or Frozen/Thawed cycles.

DETAILED DESCRIPTION:
It has been suggested that local injury to the endometrium doubles the rate of implantation and successful pregnancies in IVF patients.

Purpose

1. To determine whether performing curettage the month prior to embryo transfer (ET) increases the chance of embryo implantation.
2. To study molecular attributes of the endometrium taken at curettage and to compare them to those cycles resulting in pregnancy and those which do not result in pregnancy.

Samples will be grown as primary culture in the research laboratory and possible molecular markers and attachment assays for endometrial receptivity will be studied.

Patient selection: Patients undergoing IVF or IVF-ICSI at Ha'Emek medical center/ IVF unit. Woman over 35 years of age will be excluded since implantation failure is more likely to be due to genetic, chromosomal or cytoplasmic aberrations in their oocytes.

Proposed protocol:

1. Informed consent obtained from prospective candidates.
2. Participants randomly divided to three groups

   1. Control group
   2. Hysteroscopy and curettage performed on days 15-17 of menstrual cycle
   3. Hysteroscopy and curettage performed on days 19-22 of menstrual cycle
3. After the following menses an IVF, IVF-ICSI, or frozen embryo cycle is performed according to the unit's standard protocols.
4. The primary end point of the study will be the implantation rate after ET and the expression of possible molecular markers for endometrial receptivity in the pregnant patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* In-vitro fertilization candidate
* Normal blood coagulation

Exclusion Criteria:

* Anemia (hemoglobin under 10 mg/dl)
* Abnormal maternal karyotype
* Thrombocytopenia under 140,000
* Any contraindication to hysteroscopy or in-vitro fertilization

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-12

PRIMARY OUTCOMES:
Implantation rate
Pregnancy rate
Endometrial receptivity

CONTACTS AND LOCATIONS:
Overall Officials: Joel Geslevich, MD, Principal Investigator — haemek medical center; Eliezer Shalev, Study Chair — HaEmek Medicak Center and Technion, Israel Institute of Technology; Shlomit Goldman, Study Director — haemek medical center
Locations (1):
- Department of Obstetrics and gynecology, HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Result] La Sala GB, Montanari R, Dessanti L, Cigarini C, Sartori F. The role of diagnostic hysteroscopy and endometrial biopsy in assisted reproductive technologies. Fertil Steril. 1998 Aug;70(2):378-80. doi: 10.1016/s0015-0282(98)00147-2. PMID 9696242
- [Result] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877